CLINICAL TRIAL: NCT06108674
Title: Evaluation of the Effectiveness of Telepharmacy on Clinical Outcomes of Patients With Arterial Hypertension: Celeste Randomized Clinical Trial
Brief Title: Telepharmacy on Patients With Arterial Hypertension
Acronym: CELESTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Márcio Galvão Guimarães de Oliveira, Adjunct Professor, Federal University of Bahia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CELESTE2023
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Hypertension
Keywords: pharmaceutical care; telepharmacy; elderly patients
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telepharmacy (Experimental): Pharmaceutical care via telepharmacy
  Interventions: Other: Pharmaceutical care via telepharmacy and usual care
- In-person (Active Comparator): In-person pharmaceutical care
  Interventions: Other: Pharmaceutical care in-person and usual care

INTERVENTIONS:
Other: Pharmaceutical care via telepharmacy and usual care — Pharmacotherapeutic monitoring via telephone consultation
  Arms: Telepharmacy
Other: Pharmaceutical care in-person and usual care — Face-to-face pharmacotherapeutic monitoring
  Arms: In-person

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of a pharmaceutical care protocol via teleconsultation in the management of uncontrolled hypertension with pharmaceutical care carried out in elderly patients assisted in primary health care. The main questions it aims to answer are:

1. How effective is a pharmaceutical care protocol via teleconsultation on the clinical outcomes of elderly people with uncontrolled hypertension, when compared to in-person pharmaceutical care?
2. How effective is a pharmaceutical care protocol via teleconsultation in adherence to the treatment of elderly people with hypertension, when compared to in-person pharmaceutical care?

Participants will undergo four visits. Two visits will be for the application of instruments and measurement of clinical parameters to be carried out at the beginning and end of follow-up (visits 1 and 4). These will be carried out in a pharmacist's office at the pharmacy by previously trained pharmacists and pharmacy students. Visits 2 and 3 will be pharmaceutical consultations to be carried out in person and/or via telepharmacy.

Researchers will compare pharmaceutical care via telepharmacy with in-person pharmaceutical care to see how effective these services are in controlling blood pressure in elderly patients with uncontrolled blood pressure.

DETAILED DESCRIPTION:
Specific objectives

* Characterize the clinical and socio-demographic profile of the studied population.
* Compare the acceptance and clinical importance of interventions carried out by the pharmacist between the telepharmacy and in-person (control) groups.
* Evaluate patient adherence to medication treatment in the teleconsultation group and in person
* Evaluate patient satisfaction in the teleconsultation group and in-person consultation.
* Compare satisfaction between the telepharmacy and in-person (control) groups.

ELIGIBILITY:
Inclusion Criteria:

* Elderly patients admitted to the service with a diagnosis of systemic arterial hypertension made by a physician based on a patient report, report or medical prescription.
* Patients who present uncontrolled blood pressure at the time of assessment based on the average of three measurements using a standardized protocol at the pharmacy will be included;
* Patients must have a cell phone and know how to use it;
* Patient not have previously received pharmaceutical care.

Exclusion Criteria:

* Elderly people who are unable to use their cell phones due to cognitive impairments (Mini Mental State Examination (MMSE).
* Elderly person considered unable of using a telephone (Instrumental Activities of Daily Living)
* Elderly with controlled blood pressure according to home monitoring.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Controlling blood pressure | 3 months
  Rate of patients reaching the blood pressure target for healthy elderly people: systolic pressure of 130-139 mmHg and diastolic pressure of 70-79 mmHg; and for frail elderly people: systolic pressure of 140-149 mmHg and diastolic pressure of 70-79mmHg according to guidelines from the Brazilian Society of Cardiology of 2020

SECONDARY OUTCOMES:
Adherence to the treatment | 3 months
  Patients who score higher than eight points on the adherence scale will be considered to have high adherence, those who score between six and seven points will be classified as medium adherence and those who score less than 6 points will be classified as low adherence.
Patient satisfaction | 3 months
  The score will be calculated by the sum of the user's answers divided by the number of corresponding questions. Thus, the closer to 5, the greater the satisfaction with the service and the closer to 1, the greater the dissatisfaction.
Level of clinical significance of interventions | 3 months
  Clinical significance of the intervention as described by the DOCUMENT, which classifies interventions into four levels of clinical significance: low; light; moderate and high.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriella F Magalhães, Study Chair — UFOB; Márcio Galvão Guimarães de Oliveira, Principal Investigator — UFBA; Igor Matheus de novais Silva, Study Chair — UFBA
Locations (1):
- Farmácia Escola da UFBA, campus Anísio Teixeira, Vitória da Conquista, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Afreen N, Padilla-Tolentino E, McGinnis B. Identifying Potential High-Risk Medication Errors Using Telepharmacy and a Web-Based Survey Tool. Innov Pharm. 2021 Feb 12;12(1):10.24926/iip.v12i1.3377. doi: 10.24926/iip.v12i1.3377. eCollection 2021. PMID 34007681
- [Background] Alexander E, Butler CD, Darr A, Jenkins MT, Long RD, Shipman CJ, Stratton TP. ASHP Statement on Telepharmacy. Am J Health Syst Pharm. 2017 May 1;74(9):e236-e241. doi: 10.2146/ajhp170039. No abstract available. PMID 28438829
- [Background] Amkreutz J, Lenssen R, Marx G, Deisz R, Eisert A. Medication safety in a German telemedicine centre: Implementation of a telepharmaceutical expert consultation in addition to existing tele-intensive care unit services. J Telemed Telecare. 2020 Jan-Feb;26(1-2):105-112. doi: 10.1177/1357633X18799796. Epub 2018 Sep 25. PMID 30253681
- [Background] Ekeland AG, Bowes A, Flottorp S. Effectiveness of telemedicine: a systematic review of reviews. Int J Med Inform. 2010 Nov;79(11):736-71. doi: 10.1016/j.ijmedinf.2010.08.006. PMID 20884286
- [Background] Freeman R, Wieling W, Axelrod FB, Benditt DG, Benarroch E, Biaggioni I, Cheshire WP, Chelimsky T, Cortelli P, Gibbons CH, Goldstein DS, Hainsworth R, Hilz MJ, Jacob G, Kaufmann H, Jordan J, Lipsitz LA, Levine BD, Low PA, Mathias C, Raj SR, Robertson D, Sandroni P, Schatz I, Schondorff R, Stewart JM, van Dijk JG. Consensus statement on the definition of orthostatic hypotension, neurally mediated syncope and the postural tachycardia syndrome. Clin Auton Res. 2011 Apr;21(2):69-72. doi: 10.1007/s10286-011-0119-5. No abstract available. PMID 21431947
- [Background] Gandapur Y, Kianoush S, Kelli HM, Misra S, Urrea B, Blaha MJ, Graham G, Marvel FA, Martin SS. The role of mHealth for improving medication adherence in patients with cardiovascular disease: a systematic review. Eur Heart J Qual Care Clin Outcomes. 2016 Oct 1;2(4):237-244. doi: 10.1093/ehjqcco/qcw018. PMID 29474713
- [Background] Green BB, Cook AJ, Ralston JD, Fishman PA, Catz SL, Carlson J, Carrell D, Tyll L, Larson EB, Thompson RS. Effectiveness of home blood pressure monitoring, Web communication, and pharmacist care on hypertension control: a randomized controlled trial. JAMA. 2008 Jun 25;299(24):2857-67. doi: 10.1001/jama.299.24.2857. PMID 18577730
- [Background] Al Hamid A, Ghaleb M, Aljadhey H, Aslanpour Z. A systematic review of qualitative research on the contributory factors leading to medicine-related problems from the perspectives of adult patients with cardiovascular diseases and diabetes mellitus. BMJ Open. 2014 Sep 19;4(9):e005992. doi: 10.1136/bmjopen-2014-005992. PMID 25239295
- [Background] Diedrich L, Dockweiler C. Video-based teleconsultations in pharmaceutical care - A systematic review. Res Social Adm Pharm. 2021 Sep;17(9):1523-1531. doi: 10.1016/j.sapharm.2020.12.002. Epub 2020 Dec 13. PMID 33341405
- [Background] Margolis KL, Asche SE, Bergdall AR, Dehmer SP, Groen SE, Kadrmas HM, Kerby TJ, Klotzle KJ, Maciosek MV, Michels RD, O'Connor PJ, Pritchard RA, Sekenski JL, Sperl-Hillen JM, Trower NK. Effect of home blood pressure telemonitoring and pharmacist management on blood pressure control: a cluster randomized clinical trial. JAMA. 2013 Jul 3;310(1):46-56. doi: 10.1001/jama.2013.6549. PMID 23821088
- [Background] Williams M, Peterson GM, Tenni PC, Bindoff IK, Stafford AC. DOCUMENT: a system for classifying drug-related problems in community pharmacy. Int J Clin Pharm. 2012 Feb;34(1):43-52. doi: 10.1007/s11096-011-9583-1. Epub 2011 Nov 19. PMID 22101425
- See also: Diretrizes Brasileiras de Hipertensão Arterial - 2020. Arq Bras Cardiol. — https://abccardiol.org/wp-content/plugins/xml-to-html/include/lens/index.php?xml=0066-782X-abc-116-03-0516.xml&lang=pt-br
- See also: PORTARIA GM/MS Nº 1.348, DE 2 DE JUNHO DE 2022 — http://bvsms.saude.gov.br/bvs/saudelegis/gm/2022/prt1348_03_06_2022.html
- See also: BRASIL, Ministério da Saúde. O que é Prontuário Eletrônico do Cidadão? — http://aps.saude.gov.br/noticia/2300
- See also: Vigitel Brasil 2014: vigilância de fatores de risco e proteção para doenças crônicas por inquérito telefônico. — http://bvsms.saude.gov.br/bvs/publicacoes/vigitel_brasil_2014.pdf
- See also: Telepharmacy shows it worth in Cancer Setting. — http://www.pharmacypracticenews.com/Pharmacy-Technology-Report/Article/09-15/Telepharmacy-Shows-Its-Worth-in-Cancer-Setting/33442
- See also: Patient satisfaction with pharmacy services: translation and validation of the Pharmacy Services Questionnaire for Brazil — http://doi.org/10.1590/S0102-311X2009000100009
- See also: ORGANIZATION OF THE TELE-PHARMACEUTICAL CARE SERVICE AS AN EMERGING IN THE FIGHT AGAINST COVID-19 IN RIO GRANDE DO SUL — http://www.scielo.br/j/read/a/HxkCrtpx6qkCt7JWzgT4Yxr/